CLINICAL TRIAL: NCT05281198
Title: Effects of Exercise & Tart Cherry Ingestion on Heat Acclimation and Gut Microbiome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment of participants
Sponsor: Ohio University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 21-F-33
Record Dates: First submitted 2022-02-14; First posted 2022-03-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Heat Acclimation and Thermotolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: tart cherry (Experimental): dietary supplement: tart cherry juice
  Interventions: Dietary Supplement: tart cherry juice
- Placebo (Placebo Comparator): dietary supplement: placebo juice
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: tart cherry juice — 2, 8oz bottles of Montmorency tart cherry juice daily; 8oz taken in AM, 8oz taken in PM
  Arms: Experimental: tart cherry
Dietary Supplement: Placebo — 2, 8oz bottles of placebo juice daily; 8oz taken in AM, 8oz taken in PM
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether tart cherry supplementation effects thermotolerance and heat acclimation in human subjects exposed to exercise/heat stress.

Specific Aim I. To determine if tart cherry in combination with repeated bouts of thermally stressful exercise will impact the gut microbiome & inflammation measured via stool sample & blood samples for plasma endotoxin, inflammatory cytokines and HSP.

Specific Aim II. To determine whether whole body hyperthermia causes changes in bacterial populations in the gut microbiome, and if these changes are affected by washout or re-acclimation.

Specific Aim III. To determine whether tart cherry supplementation suppresses the ability of human subjects to acclimate to exercise/heat stress. This will be assessed via body temperature, heart rate, sweat and plasma volume responses, and exercise performance during standardized heat tolerance tests.

DETAILED DESCRIPTION:
10 recreationally trained cyclists will be recruited and will complete the study in counter-balanced randomized order (5 will start with placebo and 5 will start with tart cherry juice, then have a 4 week washout and complete the other intervention). Participants will complete 15 total sessions in the exercise physiology lab including: a VO2max test, 4 heat stress tests (pre- and post-acclimation) and 5 consecutive days of heat acclimation sessions (twice).

The VO2max test will be an incremental cycling test, starting at 80 Watts and increasing 25 Watts per minute until fatigue. The maximal Wattage will be used to determine exercise intensity during the heat stress test and heat acclimation sessions.

The heat stress test and heat acclimation sessions will occur in a controlled environment of 38C and 25% humidity. Airflow will be provided with a fan at 1 m/s. Prior to entering the controlled environment, participants will provide a mid-stream urine sample to assess hydration status via urine specific gravity (USG) and osmolality (Vapro, ELITech), then empty their bladder, measure their nude body mass on a scale (in a private bathroom in the lab), and self-insert a rectal thermometer 10cm past the anal sphincter. If the participant is dehydrated, they will be instructed to drink 500 ml of water and wait to start exercise until their hydration level is normal (USG<1.020, urine osmolality 500 800 mOsm). Researchers will then affix skin temperature sensors to the participants chest, arm, thigh, and calf and a heart rate monitor to their chest. Participants will the enter the heat chamber and sit on the bicycle for 5 minutes to get acclimated to the environment and to obtain resting levels of thermal sensation and perceived effort. Following these 5 minutes, the participant will commence exercise (described below). Participants will be provided water kept in the controlled environment (to avoid cooling) to consume ad libitum throughout all exercise sessions. Following the exercise session, participants will exit the controlled environment and void their bladder, collecting all urine in a cylinder and towel dry and assess their nude body mass. These will be used along with volume of water consumed during exercise to assess body mass changes and sweat rate.

Heat stress test:

The heat stress test will consist of cycling at 40% of their maximal Watt output for 45 minutes, followed by a 5k time trial, where they will cover the 5k in as fast a time as possible.

Heat acclimation sessions Heat acclimation sessions will be 60 minutes and will utilize an isothermic heat acclimation modality where individuals will exercise at a self-selected cadence to reach a core temperature of 38.5C. Once 38.5C has been reached, they will stop exercising and rest. Typical time to reach a core body temperature of 38.5C is 30-50 minutes, so the individual will exercise for this time, and rest for the remainder of the 60 minutes. During this rest time, body temperature will continue to rise because of metabolic heat and heat produced from exercises. However if their temperature reduces below 38.5C, they will begin exercise again to maintain temperature above 38.5C. These sessions will occur daily for 5 days.

Supplementation Participants will begin supplementation 24 hours prior to their first heat stress test and throughout their heat acclimation sessions until the final heat stress test has been completed (7 days of supplementation total). Supplementation will consist of consuming an 8 oz bottle of tart cherry juice or placebo twice daily, once in the morning and once in the evening, at least 2 hours before bed. Following a 4 week washout period, participants will complete the opposite condition (placebo or polyphenol).

The investigators will assess the impact of hyperthermia on the gut microbiome before and after heat acclimation. Participants will provide a stool sample at pre-supplementation and 24 hours post each of the heat stress tests (pre- and post-acclimation) for each of the interventions (tart cherry and placebo). Participants will collect a stool sample using a toilet hat and aliquot three small samples. They will be provided with a toilet hat, a pair of gloves, a sterile spatula, and three sterile eppendorf tubes. They will be asked to put approximately a nickle sized sample in each of these tubes. These will be placed in the freezer and brought to the lab on ice (they will be provided with a biohazard cooler bag and ice pack for transport), where they will be stored at -80C until analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-55 years old
* Recreational cyclists (>150 minutes per week of cycling exercise)
* VO2max >60th percentile according to ACSM

Exclusion Criteria:

* Previous episode of heat illness, such as heat syncope, heat exhaustion or heat stroke
* Known cardiopulmonary disease, metabolic disorders, Parkinsons Disease, or multiple sclerosis or other autonomic nervous system conditions
* diagnosed with or being treated for arthritis or any inflammatory condition (such as Lupus, gout, or Sjogrens syndrome)
* Known or suspected orthostatic hypotension or low blood pressure
* Known issues with cooling or sweating
* currently smoke or quit smoking less than one year ago
* not willing to self-insert a flexible, thin (3 mm) vinyl rectal probe and maintain this position throughout all exercise sessions.
* not willing to have blood drawn pre-supplementation and 4 times during heat stress test trials (a total of 10 times during the study).
* not willing to provide a stool sample pre- and post-heat stress tests (4 total samples).
* allergy to cherries or food dyes

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male
Enrollment: 4 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Plasma TNF-a | pre, 1 hour post heat tolerance test
  Plasma TNF-a changes from pre to 1 hour post heat tolerance test
Change in Plasma IL-6 | pre, 1 hour post heat tolerance test
  Plasma IL-6 changes from pre to 1 hour post heat tolerance test
Change in Plasma HSP70 | pre, 1 hour post heat tolerance test
  Plasma HSP70 changes from pre to 1 hour post heat tolerance test
Change in Plasma melatonin content | pre- heat tolerance test 1 (before study onset) and 2 (day 6 of exercise/heat stress)
  Plasma melatonin content from pre to post supplementation
Change in Core temperature response to heat tolerance test | heat tolerance test 1 (before study onset) and 2 (day 6 of exercise/heat stress)
  Core temperature response to heat tolerance test 1 (before study onset) and 2 (day 6 of exercise/heat stress
Change in Skin temperature response to heat tolerance test | heat tolerance test 1 (before study onset) and 2 (day 6 of exercise/heat stress)
  Skin temperature response to heat tolerance test 1 (before study onset) and 2 (day 6 of exercise/heat stress
Change in Mean body temperature response to heat tolerance test | heat tolerance test 1 (before study onset) and 2 (day 6 of exercise/heat stress)
  Mean body temperature response to heat tolerance test 1 (before study onset) and 2 (day 6 of exercise/heat stress
Change in Heart rate response to heat tolerance test | heat tolerance test 1 (before study onset) and 2 (day 6 of exercise/heat stress)
  Heart rate response to heat tolerance test 1 (before study onset) and 2 (day 6 of exercise/heat stress
Change in Physiological strain response to heat tolerance test | heat tolerance test 1 (before study onset) and 2 (day 6 of exercise/heat stress)
  Physiological strain response to heat tolerance test 1 (before study onset) and 2 (day 6 of exercise/heat stress
Change in gut microbial content | pre- heat tolerance test 1 (before study onset) and 2 (day 6 of exercise/heat stress)
  Gut microbial content from pre to post supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hillman, PhD, Principal Investigator — Division of Exercise Physiology
Locations (1):
- Ohio University Exercise Physiology Lab, Athens, Ohio, United States